CLINICAL TRIAL: NCT06582069
Title: Bleaching Effect of Solo and Combined Kiwi Extract and Ozone and Their Impact on Enamel
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mona Bedier El Lakanay, Teaching Assistant, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24/3/2024
Record Dates: First submitted 2024-08-24; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Discoloration, Tooth
MeSH Terms: conditions — Tooth Discoloration | interventions — Tooth Bleaching

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- bleaching with 2% kiwi extract. (Experimental): The fresh pulpy kiwi will be bought 200 gm of kiwi fruits were cleaned, cut into round shapes and blended with 15 mL of distilled water in a blender to obtain about 50 mL of kiwi concentrate.
  This concentrate will be filtered and then transferred into a cooling centrifuge to be processed at 2000 rpm for about 20 minutes at a temperature of 40°C.
  The extract thus collected will be stored at 4°C till further use.
  Interventions: Device: Bleaching
- bleaching using 2,350 ppm ozone gas. (Experimental): A 2,350 ppm ozone concentration at a 615 cc per minute flow rate will be supplied by a well-known ozone producing machine.
  The ppm of ozone supplied will be verified via an ozone detection device, and the ozone flow rate will be verified by a flow meter directly before the start of the experiment.
  Ozone gas will be distributed to the tooth surfaces through special trays to assure a perfect seal to prevent any ozone leakage and to be safely employed to humans
  Interventions: Device: Bleaching
- bleaching with 2% kiwi extract followed By 2,350 ppm ozone gas. (Experimental): The fresh pulpy kiwi will be bought 200 gm of kiwi fruits were cleaned, cut into round shapes and blended with 15 mL of distilled water in a blender to obtain about 50 mL of kiwi concentrate.
  This concentrate will be filtered and then transferred into a cooling centrifuge to be processed at 2000 rpm for about 20 minutes at a temperature of 40°C.
  The extract thus collected will be stored at 4°C till further use. A 2,350 ppm ozone concentration at a 615 cc per minute flow rate will be supplied by a well-known ozone producing machine.
  The ppm of ozone supplied will be verified via an ozone detection device, and the ozone flow rate will be verified by a flow meter directly before the start of the experiment.
  Ozone gas will be distributed to the tooth surfaces through special trays to assure a perfect seal to prevent any ozone leakage and to be safely employed to humans.
  Interventions: Device: Bleaching
- bleaching with 38% hydrogen peroxide. (Experimental): Application of 38% H2O2 gel for 20 minutes. Then, the H2O2 gel will be removed, and teeth will be sprayed for 10 seconds with water from a 3-in-1 syringe
  Interventions: Device: Bleaching

INTERVENTIONS:
Device: Bleaching — Bleaching

SUMMARY:
ozone therapy has been extensively used in dentistry to manage wounds healing, dental caries, oral lichen planus, gingivitis and periodontitis, halitosis, osteonecrosis of the jaw, post-surgical pain, plaque and biofilms, root canal treatment, dentin hypersensitivity, tempro-mandibular joint disorders and teeth whitening, And based on the above, in this study kiwi extract and ozone gas will be used individually and combined to evaluate the resultant effects on bleaching, enamel microhardness and micromorphology.

ELIGIBILITY:
Inclusion Criteria:

* A total of the 40 participants aged between (18-35 years) with no gender prediction.
* The participation will be entirely voluntary, and a signed statement of informed consent will be obtained prior to the start of the study.
* Systemically healthy subject based on medical and drug histories, a subject requiring scaling and polishing with moderate calculus with at least two non-adjacent hypersensitive teeth with Schiff scale scores >1 with air blast stimulus.
* Access to sound maxillary anterior teeth.
* Vitapan classical shades should be A3 or darker and lighter shades are not included.

Exclusion Criteria:

* Participants with poor oral hygiene.
* Participants with missing anterior teeth.
* Participants with unrealistic expectations.
* Participants with dental caries, those undergoing orthodontic treatment.
* Participants with a history of periodontal treatment, pregnant or lactating women and individuals with a history of asthma.
* Those who are allergic to kiwi or ozone skin therapy were excluded from the study.
* Smokers are excluded from the present study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Color change assessment | 24 Hours
  all participants will be requested to return after 24 hours to permit rehydration of tooth surfaces before shade assessment Tooth Shades will then record using colorimeter. The color change (ΔE) will be calculated using the formula: ΔE= {(ΔL) 2+ (Δa) 2+ (Δb)
Color change assessment | one month
  all participants will be requested to return after one month for tooth shades recording using colorimeter. The color change (ΔE) will be calculated using the formula: ΔE= {(ΔL) 2+ (Δa) 2+ (Δb) at one month
Color change assessment | three month
  all participants will be requested to return after one month for tooth shades recording using colorimeter. The color change (ΔE) will be calculated using the formula: ΔE= {(ΔL) 2+ (Δa) 2+ (Δb) at three months
Color change assessment | six months
  all participants will be requested to return after one month for tooth shades recording using colorimeter. The color change (ΔE) will be calculated using the formula: ΔE= {(ΔL) 2+ (Δa) 2+ (Δb) at six months

IPD SHARING:
Plan to Share IPD: Undecided